CLINICAL TRIAL: NCT04417517
Title: A Phase 1/2 Study of Evorpacept (ALX148) in Combination With Azacitidine in Patients With Higher Risk Myelodysplastic Syndrome (MDS) (ASPEN-02)
Brief Title: A Study of Evorpacept (ALX148) With Azacitidine for Higher Risk Myelodysplastic Syndrome (ASPEN-02)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: While intended to be a Phase 1/2 clinical study, the study did not proceed to Phase 2.
Sponsor: ALX Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT148002
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Higher Risk Myelodysplastic Syndromes
Keywords: ALX148; MDS; CD47; Azacitidine; HMA; SIRP-alpha; evorpacept; High risk
MeSH Terms: interventions — ALX148; Azacitidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- evorpacept (ALX148) + azacitidine (Experimental): Phase 1: Participants will receive escalating doses of evorpacept (ALX148) in combination with azacitidine 75 mg/m2 IV or subcutaneous daily for 7 days of a 28 day cycle
  Phase 2: Participants will receive evorpacept (ALX148) at the recommended Phase 2 dose in combination with azacitidine 75 mg/m2 IV or subcutaneous daily for 7 days of a 28-day cycle
  Interventions: Drug: evorpacept; Drug: azacitidine
- azacitidine (Active Comparator): Phase 2 only: Participants will receive azacitidine 75 mg/m2 IV or subcutaneous daily for 7 days of a 28-day cycle
  Interventions: Drug: azacitidine

INTERVENTIONS:
Drug: evorpacept — Fusion protein that blocks CD47-SIRPalpha pathway
  Other Names: ALX148
  Arms: evorpacept (ALX148) + azacitidine
Drug: azacitidine — Hypomethylating agent (HMA)
  Other Names: Vidaza

SUMMARY:
This Phase 1/2 clinical study will evaluate evorpacept (ALX148) in combination with azacitidine for the treatment of patients with higher risk myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
The Phase 1 will consist of a dose escalation of evorpacept (ALX148) in combination with azacitidine to evaluate safety and tolerability, and to identify the recommended Phase 2 dose of ALX148 in combination with azacitidine. The Phase 2 will evaluate the efficacy of evorpacept (ALX148) in combination with azacitidine compared to azacitidine alone for patients with previously untreated higher risk MDS.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: Diagnosis of higher risk MDS that is either previously untreated or relapsed/refractory.
* Phase 2: Diagnosis of higher risk MDS that is previously untreated.
* Adequate renal and liver function.
* Age ≥18 years.
* Adequate performance status.

Exclusion Criteria:

* Previous allogeneic hematopoietic stem cell transplant (allo-HSCT) for MDS or AML.
* Prior treatment with any anti-CD47 or anti-SIRPα (signal regulatory protein alpha) agent.
* Known active viral infections, including hepatitis B and C, human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS) related illness, or SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Phase 1: Dose Limiting Toxicities (DLT) | Up to 28 days
  Number of participants with a DLT
Phase 1: Recommended Phase 2 Dose (RP2D) | Approximately 2 years
  To identify the RP2D of ALX148 in combination with AZA
Phase 2: Complete response rate (CRR) | Approximately 6 months
  Number of participants achieving a complete response per International Working Group (IWG) criteria

CONTACTS AND LOCATIONS:
Locations (19):
- United States (10):
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - IU Simon Cancer Center, Indianapolis, Indiana
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- South Korea (5):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (4):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No